CLINICAL TRIAL: NCT06757049
Title: Clinical Outcomes of Edwards Lifesciences MITRIS RESLILA Mitral Valve in the Asian Population(THE KOREA MITRIS REGISTRY)
Brief Title: Clinical Outcomes of Edwards Lifesciences MITRIS RESLILA Mitral Valve in the Asian Population
Acronym: KOREA MITRIS
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, HO JIN KIM, Associate Professor, Asan Medical Center
Other Study IDs: 2024-1268
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Mitral Valve Insufficiency
Keywords: Mitral Valve Replacement
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate the early and mid-term safety and performance of the MITRIS RESILIA mitral valve in Asian patients in a real-world setting

DETAILED DESCRIPTION:
This study is a prospective, investigator-Investigator initiated, multicenter observational study that aims to competitively register 200 patients who have undergone mitral valve replacement surgery with the MITRIS RESILIA mitral valve at participating institutions to collect real clinical outcomes.

This study will collect data on clinical outcomes obtained during standard care for patients who undergo mitral valve replacement surgery using the MITRIS RESILIA mitral valve in South Korea.

The aim is to recruit 200 patients using the MITRIS RESILIA mitral valve (competitive recruitment, no more than 100 per institution) over a period of two years.

All patients registered in the registry will be followed for five years. Follow-up assessments will occur at 6 months, 1 year, 2 years, 3 years, and 5 years post-surgery. Including the 2-year registration period and 5 years of follow-up for result analysis, the total study duration is expected to be approximately 7.5 years. However, the overall duration may vary depending on the rate of participant registration.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 or older
2. Requires mitral valve replacement due to mitral valve dysfunction
3. The participant or their guardian can provide a written consent form approved by the IRB and agree to the research protocol and clinical follow-up schedule.

Exclusion Criteria:

1. Life expectancy of less than one year due to causes other than cardiovascular disease
2. High-risk candidates for mitral valve replacement: Society of Thoracic Surgeons Predicted Risk of Mortality 10% or greater; EuroSCORE 10% or greater; estimated surgical mortality rate by the surgeon 10% or greater
3. Chronic kidney disease: eGFR <30 mL/min/1.73m²
4. Undergoing surgery for infective endocarditis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian(REPUBLIC OF KOREA)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death | 1 year post-surgery
  death that results from a disease of the heart or blood vessels
Valve-related intervention | 1 year post-surgery
  a procedure to repair or replace a diseased or faulty heart valve
Structural valve deterioration and non-structural valve dysfunction | 1 year post-surgery
  abnormality that's not intrinsic to the valve

SECONDARY OUTCOMES:
Peak and mean trans-mitral valve pressure gradient and effective orifice area | 6 month,1 year,2 year,3 year, 5year post-surgery
  echocardiographic parameters used to assess mitral valve disease
All-cause death | 6 month,1 year,2 year,3 year, 5year post-surgery
  the total number of deaths from any cause in a given population over a specific period of time
cardiovascular death | 6 month,1 year,2 year,3 year, 5year post-surgery
  a death that results from a disease of the heart or blood vessels
Valve-related death | 6 month,1 year,2 year,3 year, 5year post-surgery
  any death that is caused by Structural valve deterioration,Nonstructural dysfunction,Valve thrombosis,Embolism,Bleeding event,Operated valve endocarditis,Death related to reintervention on the operated valve
Stroke (ischemic or hemorrhagic) | 6 month,1 year,2 year,3 year, 5year post-surgery
  a medical emergency that occurs when blood flow to the brain is blocked or a blood vessel in the brain bursts
Hospitalization due to cardiovascular disease | 6 month,1 year,2 year,3 year, 5year post-surgery
  a hospital admission with a defined cardiovascular cause
Bleeding | 6 month,1 year,2 year,3 year, 5year post-surgery
  BARC classification use.(A standardized tool for defining and categorizing bleeding events in clinical trials.)
Infective endocarditis related to the mitral valve | 6 month,1 year,2 year,3 year, 5year post-surgery
  a bacterial, viral, or fungal infection of the mitral valve leaflets
Valve-related reintervention | 6 month,1 year,2 year,3 year, 5year post-surgery
  any invasive procedure performed on the aortic valve, coronary button, or proximal aorta
Structural valve deterioration or non-structural valve dysfunction | 6 month,1 year,2 year,3 year, 5year post-surgery
  a type of valve dysfunction that involves permanent damage to the valve
Valve thrombosis | 6 month,1 year,2 year,3 year, 5year post-surgery
  a rare but life-threatening condition that occurs when a thrombus forms on a prosthetic heart valve and interferes with blood flow or valve function

CONTACTS AND LOCATIONS:
Overall Officials: HOJIN KIM, PI, Study Chair — cadiovascularthoracic surgery
Locations (1):
- Asan Medical Center, Seoul, SONGPA-GU, South Korea

IPD SHARING:
Plan to Share IPD: No